CLINICAL TRIAL: NCT00960245
Title: A Relative Bioavailability Study of Nadolol (1 x 80 mg) Tablets Under Fasting Conditions.
Brief Title: Relative Bioavailability Study of Nadolol (1 x 80 mg) Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRACS P94-102
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-08

CONDITIONS: High Blood Pressure; Migraine Headaches; Chest Pain
MeSH Terms: conditions — Hypertension; Migraine Disorders; Chest Pain | interventions — Nadolol

ARMS (2):
- 1 (Experimental): Nadolol (1 x 80 mg) Tablets (Invamed, Inc)
  Interventions: Drug: Nadolol (1 x 80 mg) Tablets (Invamed, Inc)
- 2 (Active Comparator): Corgard (1 x 80 mg) Tablets (Bristol Laboratories)
  Interventions: Drug: Corgard (1 x 80 mg) Tablets (Bristol Laboratories)

INTERVENTIONS:
Drug: Nadolol (1 x 80 mg) Tablets (Invamed, Inc)
  Arms: 1
Drug: Corgard (1 x 80 mg) Tablets (Bristol Laboratories)
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the relative bioavailability of Nadolol (1 x 80 mg) tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 1994-07; Primary Completion 1994-07 (Actual); Study Completion 1994-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Terry L. Wolff, D.O., Principal Investigator — MeritCare Broadway Health Center